CLINICAL TRIAL: NCT02869724
Title: Divided Drug Delivery : a Way to Prevent Repeated Volutary Drug Intoxications.
Brief Title: Divided Drug Delivery
Acronym: DEFIMED-1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 38RC13.577
Record Dates: First submitted 2016-07-27; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-07

CONDITIONS: Hospitalized for Voluntary Drug Intoxication
Keywords: IMV : voluntary drug intoxications; Drug; Divided prescription

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weekly divided delivery (Active Comparator): Hospitalized for voluntary drug intoxications.
  Interventions: Other: Weekly divided delivery
- Monthly divided delivery (Active Comparator): Hospitalized for voluntary drug intoxications.
  Interventions: Other: Monthly divided delivery

INTERVENTIONS:
Other: Weekly divided delivery
  Arms: Weekly divided delivery
Other: Monthly divided delivery
  Arms: Monthly divided delivery

SUMMARY:
This study will evaluate the efficacy of an advice with a weekly divided drug delivery, compared to an usual monthly delivery in the prevention of voluntary drug intoxications repeated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 65 years.
* Hospitalized after a voluntary drug intoxication.
* History of two voluntary drug intoxications at least.
* Person registered for social security.
* Signed free consent.

Exclusion Criteria:

* Patients under treatment for opiate split
* Acute or chronicgoing wild.
* Cognitive problems hindering understanding of questionnaires
* Persons targeted by articles L1121-5 to L1121-8 of CSP

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Evaluate the efficacy of an advice with a weekly divided drug delivery, compared to an usual monthly delivery in the prevention of voluntary drug intoxications repeated | 6 months
  Number of cumulative voluntary drug intoxications throughout the 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Maurice Dematteis, Professor, Principal Investigator — Grenoble Hospital University
Locations (1):
- UniversityHospitalGrenoble, La Tronche, France

REFERENCES:
- [Background] Alonso J, Angermeyer MC, Bernert S, Bruffaerts R, Brugha TS, Bryson H, de Girolamo G, Graaf R, Demyttenaere K, Gasquet I, Haro JM, Katz SJ, Kessler RC, Kovess V, Lepine JP, Ormel J, Polidori G, Russo LJ, Vilagut G, Almansa J, Arbabzadeh-Bouchez S, Autonell J, Bernal M, Buist-Bouwman MA, Codony M, Domingo-Salvany A, Ferrer M, Joo SS, Martinez-Alonso M, Matschinger H, Mazzi F, Morgan Z, Morosini P, Palacin C, Romera B, Taub N, Vollebergh WA; ESEMeD/MHEDEA 2000 Investigators, European Study of the Epidemiology of Mental Disorders (ESEMeD) Project. Psychotropic drug utilization in Europe: results from the European Study of the Epidemiology of Mental Disorders (ESEMeD) project. Acta Psychiatr Scand Suppl. 2004;(420):55-64. doi: 10.1111/j.1600-0047.2004.00331.x. PMID 15128388
- [Background] Aouba, A., Péquignot, F., Camelin, L., Laurent, F., Jougla, E. La mortalité par suicide en France en 2006. Etudes et résultats. 2009 ; (702) : 1-8.
- [Background] Beck, F., Guignard, R., Du Roscoät, E., Saïas, T. Tentatives de suicide et pensées suicidaires en France en 2010. Bulletin épidémiologique hebdomadaire. 2011 ; 47-48 : 488-492.
- [Background] Camidge DR, Wood RJ, Bateman DN. The epidemiology of self-poisoning in the UK. Br J Clin Pharmacol. 2003 Dec;56(6):613-9. doi: 10.1046/j.1365-2125.2003.01910.x. PMID 14616420
- [Background] Carter GL, Clover K, Whyte IM, Dawson AH, D'Este C. Postcards from the EDge: 24-month outcomes of a randomised controlled trial for hospital-treated self-poisoning. Br J Psychiatry. 2007 Dec;191:548-53. doi: 10.1192/bjp.bp.107.038406. PMID 18055960
- [Background] Chan-Chee, C., & Jezewski-Serra, D. Hospitalisations pour tentatives de suicide entre 2004 et 2007 en France métropolitaine. Analyse du PMSI-MCO. Bulletin épidémiologique hebdomadaire. 2011 ; 47-48 : 492-496.
- [Background] Coben JH, Davis SM, Furbee PM, Sikora RD, Tillotson RD, Bossarte RM. Hospitalizations for poisoning by prescription opioids, sedatives, and tranquilizers. Am J Prev Med. 2010 May;38(5):517-24. doi: 10.1016/j.amepre.2010.01.022. PMID 20409500
- [Background] Dumesnil, S., Grandfils, N., Le Fur, P., Mizrahi, A. Mizrahi, A. Santé, Soins et protection Sociale en France en 1996. CREDES (en ligne). Novembre 1997, (consulté le 3/4/12).
- [Background] Fedyszyn IE, Harris MG, Robinson J, Edwards J, Paxton SJ. Characteristics of suicide attempts in young people undergoing treatment for first episode psychosis. Aust N Z J Psychiatry. 2011 Oct;45(10):838-45. doi: 10.3109/00048674.2011.595687. Epub 2011 Aug 23. PMID 21861593
- [Background] Florentine JB, Crane C. Suicide prevention by limiting access to methods: a review of theory and practice. Soc Sci Med. 2010 May;70(10):1626-32. doi: 10.1016/j.socscimed.2010.01.029. Epub 2010 Feb 12. PMID 20207465
- [Background] Fournet, N., Caillère, N., Fouillet, A., Caserio-Schönemann, C., Josseran, L. Le système français de surveillance sanitaire des urgences et des décès (Sur-SaUD®). Saint-Maurice : Institut de veille sanitaire : 2011. 12p.
- [Background] Gasquet I, Negre-Pages L, Fourrier A, Nachbaur G, El-Hasnaoui A, Kovess V, Lepine JP. [Psychotropic drug use and mental psychiatric disorders in France; results of the general population ESEMeD/MHEDEA 2000 epidemiological study]. Encephale. 2005 Mar-Apr;31(2):195-206. doi: 10.1016/s0013-7006(05)82386-3. French. PMID 15959446
- [Background] Hawton K, van Heeringen K. Suicide. Lancet. 2009 Apr 18;373(9672):1372-81. doi: 10.1016/S0140-6736(09)60372-X. PMID 19376453
- [Background] Hovda KE, Bjornaas MA, Skog K, Opdahl A, Drottning P, Ekeberg O, Jacobsen D. Acute poisonings treated in hospitals in Oslo: a one-year prospective study (I): pattern of poisoning. Clin Toxicol (Phila). 2008 Jan;46(1):35-41. doi: 10.1080/15563650601185969. PMID 18167035
- [Background] Kapur N, Cooper J, Hiroeh U, May C, Appleby L, House A. Emergency department management and outcome for self-poisoning: a cohort study. Gen Hosp Psychiatry. 2004 Jan-Feb;26(1):36-41. doi: 10.1016/j.genhosppsych.2003.06.002. PMID 14757301
- [Background] Lamprecht HC, Pakrasi S, Gash A, Swann AG. Deliberate self-harm in older people revisited. Int J Geriatr Psychiatry. 2005 Nov;20(11):1090-6. doi: 10.1002/gps.1404. PMID 16250080
- [Background] Large MM, Nielssen OB. Suicide in Australia: meta-analysis of rates and methods of suicide between 1988 and 2007. Med J Aust. 2010 Apr 19;192(8):432-7. doi: 10.5694/j.1326-5377.2010.tb03580.x. PMID 20402605
- [Background] Le Pont F, Letrilliart L, Massari V, Dorleans Y, Thomas G, Flahault A. Suicide and attempted suicide in France: results of a general practice sentinel network, 1999-2001. Br J Gen Pract. 2004 Apr;54(501):282-4. PMID 15113496
- [Background] Manchikanti L, Whitfield E, Pallone F. Evolution of the National All Schedules Prescription Electronic Reporting Act (NASPER): a public law for balancing treatment of pain and drug abuse and diversion. Pain Physician. 2005 Oct;8(4):335-47. PMID 16850056
- [Background] Mann JJ, Apter A, Bertolote J, Beautrais A, Currier D, Haas A, Hegerl U, Lonnqvist J, Malone K, Marusic A, Mehlum L, Patton G, Phillips M, Rutz W, Rihmer Z, Schmidtke A, Shaffer D, Silverman M, Takahashi Y, Varnik A, Wasserman D, Yip P, Hendin H. Suicide prevention strategies: a systematic review. JAMA. 2005 Oct 26;294(16):2064-74. doi: 10.1001/jama.294.16.2064. PMID 16249421
- [Background] Mateos Rodríguez, A.A, Huerta Arroyo, A., Benito Vellisca, M.A. The epidemiology of suicide attempts using drugs. Emergencias. 2007 ; 19 : 251-254.
- [Background] Mauri MC, Cerveri G, Volonteri LS, Fiorentini A, Colasanti A, Manfre S, Borghini R, Pannacciulli E. Parasuicide and drug self-poisoning: analysis of the epidemiological and clinical variables of the patients admitted to the Poisoning Treatment Centre (CAV), Niguarda General Hospital, Milan. Clin Pract Epidemiol Ment Health. 2005 Apr 28;1(1):5. doi: 10.1186/1745-0179-1-5. PMID 15967050
- [Background] Michel, G., Aquaviva, E., Aubron, V., Purper-ouakil, D. Suicides : mieux comprendre, pour prévenir avec plus d'efficacité. In : Beck F, Guilbert P, Gautier A (dir). Baromètre santé 2005. Saint-Denis : Inpes. 2007 ; 487-506.
- [Background] Mouquet, M.C., & Bellamy, V. Suicides et tentatives de suicide en France. Etudes et Résutlats. 2006 ; 488 :1-8.
- [Background] Nordentoft M. Prevention of suicide and attempted suicide in Denmark. Epidemiological studies of suicide and intervention studies in selected risk groups. Dan Med Bull. 2007 Nov;54(4):306-69. PMID 18208680
- [Background] Owens D, Horrocks J, House A. Fatal and non-fatal repetition of self-harm. Systematic review. Br J Psychiatry. 2002 Sep;181:193-9. doi: 10.1192/bjp.181.3.193. PMID 12204922
- [Background] Prescott K, Stratton R, Freyer A, Hall I, Le Jeune I. Detailed analyses of self-poisoning episodes presenting to a large regional teaching hospital in the UK. Br J Clin Pharmacol. 2009 Aug;68(2):260-8. doi: 10.1111/j.1365-2125.2009.03458.x. PMID 19694747
- [Background] Rodríguez, A.A.M., Arroyo, A.H., and Vellisca, M.A.B. (2007). The epidemiology of suicide attempts using drugs. Emergencias. 2007 ; 19 : 251-254.
- [Background] Saviuc, P., Bedry, R., Flesch, F. Epidémiologie des intoxications médicamenteuses volontaires. Médecine Thérapeutique. 1999; 5(1): 45-8.
- [Background] Staikowsky F, Theil F, Candella S. [Trends in the pharmaceutical profile of intentional drug overdoses seen in the emergency room]. Presse Med. 2005 Jul 2;34(12):842-6. doi: 10.1016/s0755-4982(05)84060-6. French. PMID 16097205
- [Background] Simoni-Wastila L, Tompkins C. Balancing diversion control and medical necessity: the case of prescription drugs with abuse potential. Subst Use Misuse. 2001 Jul-Aug;36(9-10):1275-96. doi: 10.1081/ja-100106227. PMID 11592473
- [Background] Theil, F. Evolution qualitative des médicaments incriminés dans les intoxications médicamenteuses sur une période de 10 ans. Créteil (Paris XII). 64 pages. 2007. (Thèse de médecine).
- [Background] Tournier M, Grolleau A, Cougnard A, Molimard M, Verdoux H. Factors associated with choice of psychotropic drugs used for intentional drug overdose. Eur Arch Psychiatry Clin Neurosci. 2009 Mar;259(2):86-91. doi: 10.1007/s00406-008-0839-2. Epub 2008 Sep 19. PMID 18806918
- [Background] Vaiva G, Vaiva G, Ducrocq F, Meyer P, Mathieu D, Philippe A, Libersa C, Goudemand M. Effect of telephone contact on further suicide attempts in patients discharged from an emergency department: randomised controlled study. BMJ. 2006 May 27;332(7552):1241-5. doi: 10.1136/bmj.332.7552.1241. PMID 16735333
- [Background] Vlad IA, Fatovich DM, Fenner SG, Daly FF, Soderstrom JH, Burrows SA. Patient perceptions of the potential lethality associated with deliberate self-poisoning. Emerg Med Australas. 2011 Oct;23(5):580-6. doi: 10.1111/j.1742-6723.2011.01434.x. Epub 2011 Jun 15. PMID 21995472
- See also: Soins et protection Sociale en France en 1996. CREDES — http://www.irdes.fr/Publications/Rapports1997/rap1204.pdf